CLINICAL TRIAL: NCT03786952
Title: Stress, Sex, and the Generalization of Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio Northern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Phillip Zoladz, Professor, Ohio Northern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R15MH116337-01A1 (NIH); R15MH116337 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Psychological Stress
Keywords: stress; sex; fear; generalization; cortisol; alpha-amylase; estradiol; progesterone
MeSH Terms: conditions — Stress, Psychological; Coitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Stress, immediate, males (Experimental): Stress immediately before learning in males
  Interventions: Behavioral: Stress immediately before learning in males
- Stress, delayed, males (Experimental): Stress 30 minutes before learning in males
  Interventions: Behavioral: Stress 30 minutes before learning in males
- Sham control, immediate, males (Sham Comparator): Sham control immediately before learning in males
  Interventions: Behavioral: Sham control immediately before learning in males
- Sham control, delayed, males (Sham Comparator): Sham control 30 minutes before learning in males
  Interventions: Behavioral: Sham control 30 minutes before learning in males
- Stress, immediate, females (Experimental): Stress immediately before learning in females
  Interventions: Behavioral: Stress immediately before learning in females
- Stress, delayed, females (Experimental): Stress 30 minutes before learning in females
  Interventions: Behavioral: Stress 30 minutes before learning in females
- Sham control, immediate, females (Sham Comparator): Sham control immediately before learning in females
  Interventions: Behavioral: Sham control immediately before learning in females
- Sham control, delayed, females (Sham Comparator): Sham control 30 minutes before learning in females
  Interventions: Behavioral: Sham control 30 minutes before learning in females

INTERVENTIONS:
Behavioral: Stress immediately before learning in males — Male participants will be exposed to the socially evaluated cold pressor test immediately prior to fear learning. Participants will place their dominant hand in a bath of ice cold water for up to 3 minutes. The participants will also be informed that they are being videotaped for analysis of facial expressions and be asked to stare at a camera throughout the manipulation. Immediately following the acute stressor, participants will undergo the acquisition phase of fear conditioning.
  Arms: Stress, immediate, males
Behavioral: Sham control immediately before learning in males — Male participants will be exposed to the sham control condition (no stress) immediately prior to fear learning. Participants will place their dominant hand in a bath of lukewarm water for up to 3 minutes. Immediately following the sham control condition, participants will undergo the acquisition phase of fear conditioning.
  Arms: Sham control, immediate, males
Behavioral: Stress 30 minutes before learning in males — Male participants will be exposed to the socially evaluated cold pressor test 30 minutes prior to fear learning. Participants will place their dominant hand in a bath of ice cold water for up to 3 minutes. The participants will also be informed that they are being videotaped for analysis of facial expressions and be asked to stare at a camera throughout the manipulation. Thirty minutes following the acute stressor, participants will undergo the acquisition phase of fear conditioning.
  Arms: Stress, delayed, males
Behavioral: Sham control 30 minutes before learning in males — Male participants will be exposed to the sham control condition (no stress) 30 minutes prior to fear learning. Participants will place their dominant hand in a bath of lukewarm water for up to 3 minutes. Thirty minutes following the sham control condition, participants will undergo the acquisition phase of fear conditioning.
  Arms: Sham control, delayed, males
Behavioral: Stress immediately before learning in females — Female participants will be exposed to the socially evaluated cold pressor test immediately prior to fear learning. Participants will place their dominant hand in a bath of ice cold water for up to 3 minutes. The participants will also be informed that they are being videotaped for analysis of facial expressions and be asked to stare at a camera throughout the manipulation. Immediately following the acute stressor, participants will undergo the acquisition phase of fear conditioning.
  Arms: Stress, immediate, females
Behavioral: Sham control immediately before learning in females — Female participants will be exposed to the sham control condition (no stress) immediately prior to fear learning. Participants will place their dominant hand in a bath of lukewarm water for up to 3 minutes. Immediately following the sham control condition, participants will undergo the acquisition phase of fear conditioning.
  Arms: Sham control, immediate, females
Behavioral: Stress 30 minutes before learning in females — Female participants will be exposed to the socially evaluated cold pressor test 30 minutes prior to fear learning. Participants will place their dominant hand in a bath of ice cold water for up to 3 minutes. The participants will also be informed that they are being videotaped for analysis of facial expressions and be asked to stare at a camera throughout the manipulation. Thirty minutes following the acute stressor, participants will undergo the acquisition phase of fear conditioning.
  Arms: Stress, delayed, females
Behavioral: Sham control 30 minutes before learning in females — Female participants will be exposed to the sham control condition (no stress) 30 minutes prior to fear learning. Participants will place their dominant hand in a bath of lukewarm water for up to 3 minutes. Thirty minutes following the sham control condition, participants will undergo the acquisition phase of fear conditioning.
  Arms: Sham control, delayed, females

SUMMARY:
The impact of well-known risk factors for such disorders (stress, biological sex, anxiety-related dispositions) on fear generalization will be examined. Findings from this study may provide insight into how these risk factors influence the development and/or maintenance of psychological disorders that involve overgeneralization of fear and could facilitate future approaches to their treatment.

DETAILED DESCRIPTION:
Many researchers approach the etiology of trauma-, stressor-, and anxiety-related mental disorders from the perspective of classical conditioning processes gone awry. According to this view, abnormal associative relationships between neutral, conditioned stimuli (CSs) and aversive, unconditioned stimuli (USs) underlie pathological anxiety and result in unusually intense fear memories or fear memories that cannot be properly extinguished. Recent work has expanded this view by showing that many psychological disorders involving pathological anxiety are associated with an exaggerated form of the commonly adaptive classical conditioning phenomenon, stimulus generalization, leading individuals with such disorders to respond with fear and anxiety to a variety of environmental contexts and cues that should not be threatening. Few studies have been conducted in humans to better understand the process of fear generalization, and factors that might influence susceptibility to overgeneralize fear have yet to be assessed. It is well-known that stress, biological sex, and anxiety-related dispositions of an individual increase one's susceptibility for pathological anxiety and significantly impact fear learning; thus, it is possible that such factors, alone or in combination, contribute to clinical anxiety by influencing fear generalization processes. Aim 1 of the present study is to determine the effects of acute stress and its physiological correlates on fear generalization in human participants. Because acute stress profoundly impacts cognitive brain areas that underlie generalization, it is predicted that acute stress will enhance or impair fear generalization, depending on when the stressor is administered relative to fear learning. Aim 2 is to assess the role of biological sex in fear generalization and acute stress-induced changes in such processes. Females are more likely than males to develop several psychological disorders that involve pathological anxiety, and research has consistently reported sex-related differences in fear learning and stress-induced alterations of fear learning, effects that have been associated with ovarian hormones. Thus, it is predicted that females will exhibit greater fear generalization than males that will be impacted differently by stress. It is also hypothesized that the observed effects will correlate with estradiol and progesterone in females. The final aim of this project (Aim 3) is to evaluate the relationship between childhood stress, dispositional anxiety, and fear generalization. Early life stress has been repeatedly associated with altered stress responses and the development of anxiety-related phenotypes, yet the influence of childhood stress and trait anxiety on fear generalization have yet to be examined. This study will be the first to examine how several factors that are known to increase susceptibility for trauma-, stressor, and anxiety-related psychological disorders impact fear generalization in human subjects. The resulting findings will provide important insight into the etiology of such disorders, which could aid future approaches to their treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Registered student at Ohio Northern University in Ada, Ohio

Exclusion Criteria:

* Regular use of tobacco or recreational drugs (e.g., marijuana, cocaine, heroin, etc.)
* Previous diagnosis of Raynaud's disease or peripheral vascular disease
* Previous diagnosis of skin diseases (e.g., severe psoriasis, eczema, scleroderma)
* History of syncope or vasovagal response to stress
* History of any heart conditions or cardiovascular issues (e.g., high blood pressure)
* History of severe head trauma
* Current treatment with narcotics, beta-blockers, or steroids
* Previous diagnosis of substance use disorder
* Regular nightshift work
* Hearing loss
* Consumed alcohol in past 24 hours
* Engaged in strenuous exercise in past 24 hours
* Ate or drank anything but water in past 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Zoladz, Ph.D., Principal Investigator — Ohio Northern University
Locations (1):
- Ohio Northern University, Ada, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data and data from descriptive/raw measures were submitted on a semi-annual basis to the NIMH Data Archive
Time Frame: Data were shared on a semi-annual basis, beginning in January 2020.
Access Criteria: NIMH Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Started | 56 | 59 | 58 | 57 | 97 | 87 | 94 | 98
Completed | 56 | 59 | 58 | 57 | 97 | 87 | 94 | 98
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females | Total
Number analyzed (Participants) | 56 | 59 | 58 | 57 | 97 | 87 | 94 | 98 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.38 (1.65) | 19.95 (1.79) | 19.19 (1.26) | 19.61 (1.32) | 18.77 (0.98) | 19.39 (3.06) | 18.84 (0.86) | 18.97 (1.16) | 19.19 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 97 | 87 | 94 | 98 | 376
  Male | 56 | 59 | 58 | 57 | 0 | 0 | 0 | 0 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 1 | 4 | 0 | 6 | 4 | 20
  Not Hispanic or Latino | 55 | 57 | 56 | 56 | 93 | 87 | 88 | 94 | 586
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 3 | 3 | 2 | 2 | 6 | 6 | 1 | 4 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 7 | 4 | 5 | 3 | 2 | 3 | 2 | 29
  White | 50 | 48 | 52 | 50 | 87 | 79 | 90 | 90 | 546
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 56 | 59 | 58 | 57 | 97 | 87 | 94 | 98 | 606
Height [Mean (Standard Deviation); unit: inches] | 70 (2.83645) | 70.3051 (3.07523) | 71.1724 (2.34811) | 70.5088 (3.26301) | 64.7526 (3.06197) | 65.1552 (2.92375) | 65.734 (3.05567) | 65.0332 (3.00121) | 67.1894 (3.94860)
Weight [Mean (Standard Deviation); unit: pounds] | 175.6429 (39.54810) | 175.7458 (32.51980) | 182.5862 (37.76522) | 192.8772 (44.19400) | 146.1237 (34.88889) | 149.2989 (32.93020) | 154.7553 (36.01424) | 153.4286 (41.21405) | 162.5990 (40.33790)

OUTCOME MEASURES:

1. Primary Outcome: Fear-potentiated Startle Responses to the CS+ and CS- During Acquisition
Description: Peak eyeblink startle responses 20-200 ms following presentation of a startle probe were measured. Startle responses were assessed for each of 3 trial types: (1) following the startle probe alone [noise alone (NA) trials], (2) following the CS+ and startle probe (CS+ trials), and (3) following the CS- and startle probe (CS- trials). Participants were exposed to 16 blocks of trials, and each block included 1 presentation of each trial type. During the last 12 blocks, CS+ trials also included the presentation of an aversive US. For each block, startle responses to NA trials were subtracted from startle responses to CS+ trials and from startle responses to CS- trials to create 2 separate fear-potentiated startle response measures: 1 for the CS+ and 1 for the CS-. Average fear-potentiated startle responses to the CS+ and CS- during the last 4 blocks of trials were used as an indicator of fear learning (greater responses to the CS+, relative to the CS-, indicated greater learning).
Time Frame: Average of the responses from trial block 13, trial block 14, trial block 15, and trial block 16 on Day 1
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some fear-potentiated startle responses were unable to be obtained from participants due to technical issues (e.g., poor electrode conductance).
Measure: Mean (Standard Error); unit: Fear-potentiated startle (microvolts)
Groups:
- Stress, Immediate, Males, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Stress, Delayed, Females, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: Fear-potentiated startle responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: Fear-potentiated startle responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 36 | 36 | 39 | 39 | 72 | 72 | 66 | 66 | 71 | 71 | 72 | 72
Fear-potentiated startle (microvolts) | 52.059 (9.46) | 19.162 (7.955) | 44.388 (9.46) | 9.732 (7.955) | 42.123 (9.972) | 20.215 (8.385) | 47.904 (9.581) | 26.64 (8.056) | 64.313 (7.051) | 14.437 (5.929) | 75.269 (7.365) | 33.479 (6.193) | 61.243 (7.101) | 26.584 (5.971) | 62.828 (7.051) | 21.856 (5.929)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.453, ANOVA

2. Primary Outcome: EMG Responses to CS+, CS-, and Generalization Stimuli During Generalization Testing
Description: Peak eyeblink startle responses 20-200 ms following the presentation of a startle probe were measured. Startle responses were assessed for each of 10 trial types: (1) following the startle probe alone [noise alone (NA) trials], (2) following the CS+ and startle probe (CS+ trials), (3) following each of 7 generalization stimuli and startle probe (GS trials), and (4) following the CS- and startle probe (CS- trials). Participants were exposed to 3 blocks of trials, and each block included 1 presentation of each trial type. For each block, startle responses to the NA trials were subtracted from startle responses to the CS+, GSs, and CS- trials to create separate fear-potentiated startle response measures for each of the 9 different stimuli. Average fear-potentiated startle responses to each stimulus across all 3 blocks were used as an indicator of fear expression. Greater scores for the generalization stimuli (GS) indicated a greater generalization of fear.
Time Frame: Average of responses from all trials on Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Fear-potentiated startle (microvolts)
Groups:
- Stress, Immediate, Males, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in females stressed 30 min before learning
- Sham Control, Immediate, Females, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: Fear-potentiated startle responses to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS1: Fear-potentiated startle responses to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS2: Fear-potentiated startle responses to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS3: Fear-potentiated startle responses to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS4: Fear-potentiated startle responses to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS5: Fear-potentiated startle responses to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS6: Fear-potentiated startle responses to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS7: Fear-potentiated startle responses to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: Fear-potentiated startle responses to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, GS1 | Stress, Immediate, Males, GS2 | Stress, Immediate, Males, GS3 | Stress, Immediate, Males, GS4 | Stress, Immediate, Males, GS5 | Stress, Immediate, Males, GS6 | Stress, Immediate, Males, GS7 | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, GS1 | Stress, Delayed, Males, GS2 | Stress, Delayed, Males, GS3 | Stress, Delayed, Males, GS4 | Stress, Delayed, Males, GS5 | Stress, Delayed, Males, GS6 | Stress, Delayed, Males, GS7 | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, GS1 | Sham Control, Immediate, Males, GS2 | Sham Control, Immediate, Males, GS3 | Sham Control, Immediate, Males, GS4 | Sham Control, Immediate, Males, GS5 | Sham Control, Immediate, Males, GS6 | Sham Control, Immediate, Males, GS7 | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, GS1 | Sham Control, Delayed, Males, GS2 | Sham Control, Delayed, Males, GS3 | Sham Control, Delayed, Males, GS4 | Sham Control, Delayed, Males, GS5 | Sham Control, Delayed, Males, GS6 | Sham Control, Delayed, Males, GS7 | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, GS1 | Stress, Immediate, Females, GS2 | Stress, Immediate, Females, GS3 | Stress, Immediate, Females, GS4 | Stress, Immediate, Females, GS5 | Stress, Immediate, Females, GS6 | Stress, Immediate, Females, GS7 | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, GS1 | Stress, Delayed, Females, GS2 | Stress, Delayed, Females, GS3 | Stress, Delayed, Females, GS4 | Stress, Delayed, Females, GS5 | Stress, Delayed, Females, GS6 | Stress, Delayed, Females, GS7 | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, GS1 | Sham Control, Immediate, Females, GS2 | Sham Control, Immediate, Females, GS3 | Sham Control, Immediate, Females, GS4 | Sham Control, Immediate, Females, GS5 | Sham Control, Immediate, Females, GS6 | Sham Control, Immediate, Females, GS7 | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, GS1 | Sham Control, Delayed, Females, GS2 | Sham Control, Delayed, Females, GS3 | Sham Control, Delayed, Females, GS4 | Sham Control, Delayed, Females, GS5 | Sham Control, Delayed, Females, GS6 | Sham Control, Delayed, Females, GS7 | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 42 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 73 | 73 | 73 | 73 | 73 | 73 | 73 | 73 | 73 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 76 | 76 | 76 | 76 | 76 | 76 | 76 | 76 | 76
Fear-potentiated startle (microvolts) | 52.059 (9.552) | 42.389 (8.467) | 24.461 (8.215) | 36.099 (7.563) | 25.637 (7.085) | 13.225 (7.130) | 36.013 (7.759) | 16.838 (7.797) | 19.063 (7.897) | 51.595 (9.552) | 47.292 (8.467) | 23.265 (8.215) | 26.790 (7.563) | 17.900 (7.085) | 17.642 (7.130) | 18.197 (7.759) | 17.472 (7.797) | 18.542 (7.897) | 59.295 (10.317) | 36.931 (9.146) | 29.738 (8.874) | 32.878 (8.169) | 31.296 (7.652) | 28.073 (7.701) | 32.893 (8.380) | 21.807 (8.422) | 25.547 (8.529) | 68.576 (9.668) | 52.235 (8.57) | 36.234 (8.315) | 33.031 (7.655) | 37.434 (7.171) | 22.264 (7.216) | 29.489 (7.853) | 27.508 (7.892) | 35.165 (7.993) | 59.043 (7.245) | 49.511 (6.422) | 37.996 (6.231) | 38.498 (5.737) | 32.051 (5.374) | 26.428 (5.408) | 48.603 (5.885) | 32.181 (5.914) | 19.585 (5.99) | 57.618 (7.563) | 51.025 (6.704) | 31.866 (6.505) | 36.741 (5.988) | 26.989 (5.609) | 23.399 (5.645) | 42.591 (6.143) | 25.380 (6.173) | 28.132 (6.252) | 51.693 (7.148) | 49.296 (6.336) | 29.101 (6.148) | 36.858 (5.660) | 28.705 (5.302) | 24.520 (5.335) | 37.415 (5.806) | 28.944 (5.835) | 24.180 (5.909) | 65.451 (7.101) | 61.473 (6.294) | 40.557 (6.107) | 42.141 (5.622) | 30.156 (5.267) | 34.117 (5.300) | 43.093 (5.768) | 34.696 (5.796) | 42.714 (5.870)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, GS1 vs Stress, Immediate, Males, GS2 vs Stress, Immediate, Males, GS3 vs Stress, Immediate, Males, GS4 vs Stress, Immediate, Males, GS5 vs Stress, Immediate, Males, GS6 vs Stress, Immediate, Males, GS7 vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, GS1 vs Stress, Delayed, Males, GS2 vs Stress, Delayed, Males, GS3 vs Stress, Delayed, Males, GS4 vs Stress, Delayed, Males, GS5 vs Stress, Delayed, Males, GS6 vs Stress, Delayed, Males, GS7 vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, GS1 vs Sham Control, Immediate, Males, GS2 vs Sham Control, Immediate, Males, GS3 vs Sham Control, Immediate, Males, GS4 vs Sham Control, Immediate, Males, GS5 vs Sham Control, Immediate, Males, GS6 vs Sham Control, Immediate, Males, GS7 vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, GS1 vs Sham Control, Delayed, Males, GS2 vs Sham Control, Delayed, Males, GS3 vs Sham Control, Delayed, Males, GS4 vs Sham Control, Delayed, Males, GS5 vs Sham Control, Delayed, Males, GS6 vs Sham Control, Delayed, Males, GS7 vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, GS1 vs Stress, Immediate, Females, GS2 vs Stress, Immediate, Females, GS3 vs Stress, Immediate, Females, GS4 vs Stress, Immediate, Females, GS5 vs Stress, Immediate, Females, GS6 vs Stress, Immediate, Females, GS7 vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, GS1 vs Stress, Delayed, Females, GS2 vs Stress, Delayed, Females, GS3 vs Stress, Delayed, Females, GS4 vs Stress, Delayed, Females, GS5 vs Stress, Delayed, Females, GS6 vs Stress, Delayed, Females, GS7 vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, GS1 vs Sham Control, Immediate, Females, GS2 vs Sham Control, Immediate, Females, GS3 vs Sham Control, Immediate, Females, GS4 vs Sham Control, Immediate, Females, GS5 vs Sham Control, Immediate, Females, GS6 vs Sham Control, Immediate, Females, GS7 vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, GS1 vs Sham Control, Delayed, Females, GS2 vs Sham Control, Delayed, Females, GS3 vs Sham Control, Delayed, Females, GS4 vs Sham Control, Delayed, Females, GS5 vs Sham Control, Delayed, Females, GS6 vs Sham Control, Delayed, Females, GS7 vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.931, ANOVA

3. Primary Outcome: Skin Conductance Responses to CS+ and CS- During Acquisition
Description: Electrodermal activity was measured following presentation of the CS+ and CS- during acquisition on Day 1. Participants were exposed to 16 blocks of trials, with each block including a single presentation of each stimulus. During the last 12 blocks, CS+ trials included the presentation of an aversive US. For each block, skin conductance responses were quantified by calculating the average increase in electrodermal activity (from a 1 s pre-stimulus baseline) 3-6 s after CS+ or CS- onset. Average skin conductance responses to the CS+ and CS- during the last 4 blocks of trials were used as an indicator of fear learning (greater responses to the CS+, relative to the CS-, indicated greater learning).
Time Frame: Average of the responses from trial block 13, trial block 14, trial block 15, and trial block 16 on Day 1
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some skin conductance responses were unable to be obtained from participants due to technical issues (e.g., poor electrode conductance).
Measure: Mean (Standard Error); unit: Skin conductance response (μSiemens)
Groups:
- Stress, Immediate, Males, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Stress, Delayed, Females, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: Skin conductance responses to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: Skin conductance responses to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 39 | 39 | 41 | 41 | 36 | 36 | 39 | 39 | 72 | 72 | 59 | 59 | 73 | 73 | 76 | 76
Skin conductance response (μSiemens) | .107 (.042) | .070 (.039) | .138 (.041) | .090 (.038) | .112 (.043) | .102 (.040) | .163 (.042) | .105 (.039) | .153 (.031) | .084 (.029) | .135 (.034) | .078 (.032) | .206 (.031) | .072 (.028) | .244 (.030) | .096 (.028)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.923, ANOVA

4. Primary Outcome: Skin Conductance Responses to CS+, Generalization Stimuli, and CS- During Generalization Testing
Description: Electrodermal activity was measured following presentation of the CS+, 7 generalization stimuli (GSs), and CS- during generalization testing on Day 2. Participants were exposed to 3 blocks of trials, with each block including a single presentation of each stimulus. For each block, skin conductance responses were quantified by calculating the average increase in electrodermal activity (from a 1 s pre-stimulus baseline) 3-6 s after onset of the CS+, 7 GSs, or CS- onset.. Average skin conductance responses to each stimulus across all 3 blocks were used as an indicator of fear expression. Greater scores for the generalization stimuli (GS) indicated a greater generalization of fear.
Time Frame: Average of responses from all trials on Day 2
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Skin conductance response (μSiemens)
Groups:
- Stress, Immediate, Males, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in females stressed 30 min before learning
- Sham Control, Immediate, Females, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: Skin conductance responses to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS1: Skin conductance responses to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS2: Skin conductance responses to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS3: Skin conductance responses to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS4: Skin conductance responses to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS5: Skin conductance responses to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS6: Skin conductance responses to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS7: Skin conductance responses to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: Skin conductance responses to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, GS1 | Stress, Immediate, Males, GS2 | Stress, Immediate, Males, GS3 | Stress, Immediate, Males, GS4 | Stress, Immediate, Males, GS5 | Stress, Immediate, Males, GS6 | Stress, Immediate, Males, GS7 | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, GS1 | Stress, Delayed, Males, GS2 | Stress, Delayed, Males, GS3 | Stress, Delayed, Males, GS4 | Stress, Delayed, Males, GS5 | Stress, Delayed, Males, GS6 | Stress, Delayed, Males, GS7 | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, GS1 | Sham Control, Immediate, Males, GS2 | Sham Control, Immediate, Males, GS3 | Sham Control, Immediate, Males, GS4 | Sham Control, Immediate, Males, GS5 | Sham Control, Immediate, Males, GS6 | Sham Control, Immediate, Males, GS7 | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, GS1 | Sham Control, Delayed, Males, GS2 | Sham Control, Delayed, Males, GS3 | Sham Control, Delayed, Males, GS4 | Sham Control, Delayed, Males, GS5 | Sham Control, Delayed, Males, GS6 | Sham Control, Delayed, Males, GS7 | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, GS1 | Stress, Immediate, Females, GS2 | Stress, Immediate, Females, GS3 | Stress, Immediate, Females, GS4 | Stress, Immediate, Females, GS5 | Stress, Immediate, Females, GS6 | Stress, Immediate, Females, GS7 | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, GS1 | Stress, Delayed, Females, GS2 | Stress, Delayed, Females, GS3 | Stress, Delayed, Females, GS4 | Stress, Delayed, Females, GS5 | Stress, Delayed, Females, GS6 | Stress, Delayed, Females, GS7 | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, GS1 | Sham Control, Immediate, Females, GS2 | Sham Control, Immediate, Females, GS3 | Sham Control, Immediate, Females, GS4 | Sham Control, Immediate, Females, GS5 | Sham Control, Immediate, Females, GS6 | Sham Control, Immediate, Females, GS7 | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, GS1 | Sham Control, Delayed, Females, GS2 | Sham Control, Delayed, Females, GS3 | Sham Control, Delayed, Females, GS4 | Sham Control, Delayed, Females, GS5 | Sham Control, Delayed, Females, GS6 | Sham Control, Delayed, Females, GS7 | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 37 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 57 | 57 | 57 | 57 | 57 | 57 | 57 | 57 | 57 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 67 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75
Skin conductance response (μSiemens) | .193 (.049) | .156 (.047) | .103 (.039) | .114 (.043) | .072 (.039) | .046 (.040) | .241 (.053) | .246 (.049) | .094 (.039) | .270 (.047) | .262 (.045) | .140 (.037) | .177 (.041) | .095 (.037) | .118 (.038) | .254 (.050) | .101 (.047) | .116 (.037) | .127 (.054) | .154 (.051) | .081 (.043) | .158 (.047) | .041 (.042) | .053 (.044) | .260 (.058) | .103 (.054) | .138 (.042) | .196 (.048) | .212 (.045) | .107 (.038) | .129 (.041) | .067 (.037) | .035 (.039) | .218 (.051) | .193 (.047) | .075 (.037) | .225 (.036) | .184 (.035) | .119 (.029) | .168 (.032) | .123 (.029) | .132 (.03) | .232 (.039) | .196 (.036) | .093 (.028) | .213 (.040) | .201 (.038) | .098 (.032) | .147 (.035) | .085 (.031) | .122 (.033) | .252 (.043) | .127 (.040) | .074 (.031) | .226 (.037) | .199 (.035) | .094 (.029) | .150 (.032) | .100 (.029) | .097 (.030) | .259 (.039) | .137 (.037) | .109 (.029) | .243 (.035) | .261 (.033) | .100 (.028) | .195 (.030) | .113 (.027) | .138 (.028) | .326 (.037) | .198 (.035) | .158 (.027)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, GS1 vs Stress, Immediate, Males, GS2 vs Stress, Immediate, Males, GS3 vs Stress, Immediate, Males, GS4 vs Stress, Immediate, Males, GS5 vs Stress, Immediate, Males, GS6 vs Stress, Immediate, Males, GS7 vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, GS1 vs Stress, Delayed, Males, GS2 vs Stress, Delayed, Males, GS3 vs Stress, Delayed, Males, GS4 vs Stress, Delayed, Males, GS5 vs Stress, Delayed, Males, GS6 vs Stress, Delayed, Males, GS7 vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, GS1 vs Sham Control, Immediate, Males, GS2 vs Sham Control, Immediate, Males, GS3 vs Sham Control, Immediate, Males, GS4 vs Sham Control, Immediate, Males, GS5 vs Sham Control, Immediate, Males, GS6 vs Sham Control, Immediate, Males, GS7 vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, GS1 vs Sham Control, Delayed, Males, GS2 vs Sham Control, Delayed, Males, GS3 vs Sham Control, Delayed, Males, GS4 vs Sham Control, Delayed, Males, GS5 vs Sham Control, Delayed, Males, GS6 vs Sham Control, Delayed, Males, GS7 vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, GS1 vs Stress, Immediate, Females, GS2 vs Stress, Immediate, Females, GS3 vs Stress, Immediate, Females, GS4 vs Stress, Immediate, Females, GS5 vs Stress, Immediate, Females, GS6 vs Stress, Immediate, Females, GS7 vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, GS1 vs Stress, Delayed, Females, GS2 vs Stress, Delayed, Females, GS3 vs Stress, Delayed, Females, GS4 vs Stress, Delayed, Females, GS5 vs Stress, Delayed, Females, GS6 vs Stress, Delayed, Females, GS7 vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, GS1 vs Sham Control, Immediate, Females, GS2 vs Sham Control, Immediate, Females, GS3 vs Sham Control, Immediate, Females, GS4 vs Sham Control, Immediate, Females, GS5 vs Sham Control, Immediate, Females, GS6 vs Sham Control, Immediate, Females, GS7 vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, GS1 vs Sham Control, Delayed, Females, GS2 vs Sham Control, Delayed, Females, GS3 vs Sham Control, Delayed, Females, GS4 vs Sham Control, Delayed, Females, GS5 vs Sham Control, Delayed, Females, GS6 vs Sham Control, Delayed, Females, GS7 vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.399, ANOVA

5. Primary Outcome: US Expectancy Ratings to CS+ and CS- During Acquisition
Description: Participants were exposed to 16 blocks of trials, and each block included 1 presentation of the CS+ and one presentation of the CS-. During the last 12 blocks, CS+ trials included the presentation of an aversive US. During each trial, participants pressed, within 3 seconds of stimulus onset, a button marked "+" if they expected the stimulus to be followed by the US, a button marked "-" if they did not expect the stimulus to be followed by the US, or a button marked "0" if they were uncertain. For the purpose of data analysis, + was scored as +1, - were scored as -1, and 0 was scored as 0. Average expectancy ratings during the last 4 blocks of trials were used as an indicator of fear learning (greater responses to the CS+, relative to the CS-, indicated greater learning).
Time Frame: Average of the ratings from trial block 13, trial block 14, trial block 15, and trial block 16 on Day 1
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some US expectancy ratings were unable to be obtained from participants due to technical issues (e.g., response pad malfunction) or participant error.
Measure: Mean (Standard Error); unit: score on scale from -1 to +1
Groups:
- Stress, Immediate, Males, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Stress, Delayed, Females, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: US expectancy ratings to the CS+ during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: US expectancy ratings to the CS- during the conditioning phase of acquisition on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 39 | 39 | 42 | 42 | 37 | 37 | 43 | 43 | 74 | 74 | 66 | 66 | 72 | 72 | 74 | 74
score on scale from -1 to +1 | .737 (.064) | -.865 (.068) | .964 (.062) | -.954 (.066) | .797 (.066) | -.775 (.070) | .860 (.061) | -.907 (.065) | .807 (.047) | -.782 (.050) | .867 (.050) | -.845 (.053) | .889 (.047) | -.840 (.050) | .881 (.047) | -.898 (.050)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.872, ANOVA

6. Primary Outcome: US Expectancy Ratings to CS+, CS-, and Generalization Stimuli During Generalization Testing
Description: Participants were exposed to 3 blocks of trials, and each block included 1 presentation of the CS+, one presentation of each of 7 generalization stimuli (GSs), and one presentation of the CS-. Participants were instructed to press, within 3 seconds of stimulus onset, a button marked "+" if they expected the stimulus to be followed by the US, a button marked "-" if they did not expect the stimulus to be followed by the US, or a button marked "0" if they were uncertain. For the purpose of data analysis, + was scored as +1, - was scored as -1, and 0 was scored as 0. Average expectancy ratings for each stimulus across all 3 blocks were used as an indicator of fear. Greater scores for the generalization stimuli (GS) indicated a greater generalization of fear.
Time Frame: Average of ratings from all trials on Day 2
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on scale from -1 to +1
Groups:
- Stress, Immediate, Males, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Immediate, Males, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in males stressed immediately before learning
- Stress, Delayed, Males, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in males stressed 30 min before learning
- Stress, Delayed, Males, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in males stressed 30 min before learning
- Sham Control, Immediate, Males, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Males, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Males, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Immediate, Females, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in females stressed immediately before learning
- Stress, Delayed, Females, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in females stressed 30 min before learning
- Stress, Delayed, Females, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in females stressed 30 min before learning
- Sham Control, Immediate, Females, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Immediate, Females, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females, CS+: US expectancy ratings to the CS+ during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS1: US expectancy ratings to the GS1 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS2: US expectancy ratings to the GS2 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS3: US expectancy ratings to the GS3 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS4: US expectancy ratings to the GS4 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS5: US expectancy ratings to the GS5 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS6: US expectancy ratings to the GS6 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, GS7: US expectancy ratings to the GS7 during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
- Sham Control, Delayed, Females, CS-: US expectancy ratings to the CS- during generalization testing on Day 2 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males, CS+ | Stress, Immediate, Males, GS1 | Stress, Immediate, Males, GS2 | Stress, Immediate, Males, GS3 | Stress, Immediate, Males, GS4 | Stress, Immediate, Males, GS5 | Stress, Immediate, Males, GS6 | Stress, Immediate, Males, GS7 | Stress, Immediate, Males, CS- | Stress, Delayed, Males, CS+ | Stress, Delayed, Males, GS1 | Stress, Delayed, Males, GS2 | Stress, Delayed, Males, GS3 | Stress, Delayed, Males, GS4 | Stress, Delayed, Males, GS5 | Stress, Delayed, Males, GS6 | Stress, Delayed, Males, GS7 | Stress, Delayed, Males, CS- | Sham Control, Immediate, Males, CS+ | Sham Control, Immediate, Males, GS1 | Sham Control, Immediate, Males, GS2 | Sham Control, Immediate, Males, GS3 | Sham Control, Immediate, Males, GS4 | Sham Control, Immediate, Males, GS5 | Sham Control, Immediate, Males, GS6 | Sham Control, Immediate, Males, GS7 | Sham Control, Immediate, Males, CS- | Sham Control, Delayed, Males, CS+ | Sham Control, Delayed, Males, GS1 | Sham Control, Delayed, Males, GS2 | Sham Control, Delayed, Males, GS3 | Sham Control, Delayed, Males, GS4 | Sham Control, Delayed, Males, GS5 | Sham Control, Delayed, Males, GS6 | Sham Control, Delayed, Males, GS7 | Sham Control, Delayed, Males, CS- | Stress, Immediate, Females, CS+ | Stress, Immediate, Females, GS1 | Stress, Immediate, Females, GS2 | Stress, Immediate, Females, GS3 | Stress, Immediate, Females, GS4 | Stress, Immediate, Females, GS5 | Stress, Immediate, Females, GS6 | Stress, Immediate, Females, GS7 | Stress, Immediate, Females, CS- | Stress, Delayed, Females, CS+ | Stress, Delayed, Females, GS1 | Stress, Delayed, Females, GS2 | Stress, Delayed, Females, GS3 | Stress, Delayed, Females, GS4 | Stress, Delayed, Females, GS5 | Stress, Delayed, Females, GS6 | Stress, Delayed, Females, GS7 | Stress, Delayed, Females, CS- | Sham Control, Immediate, Females, CS+ | Sham Control, Immediate, Females, GS1 | Sham Control, Immediate, Females, GS2 | Sham Control, Immediate, Females, GS3 | Sham Control, Immediate, Females, GS4 | Sham Control, Immediate, Females, GS5 | Sham Control, Immediate, Females, GS6 | Sham Control, Immediate, Females, GS7 | Sham Control, Immediate, Females, CS- | Sham Control, Delayed, Females, CS+ | Sham Control, Delayed, Females, GS1 | Sham Control, Delayed, Females, GS2 | Sham Control, Delayed, Females, GS3 | Sham Control, Delayed, Females, GS4 | Sham Control, Delayed, Females, GS5 | Sham Control, Delayed, Females, GS6 | Sham Control, Delayed, Females, GS7 | Sham Control, Delayed, Females, CS-
Number analyzed (Participants) | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 45 | 45 | 45 | 45 | 45 | 45 | 45 | 45 | 45 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 79 | 79 | 79 | 79 | 79 | 79 | 79 | 79 | 79 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 80 | 80 | 80 | 80 | 80 | 80 | 80 | 80 | 80
score on scale from -1 to +1 | .217 (.119) | .140 (.094) | -.357 (.111) | -.527 (.095) | -.822 (.069) | -.810 (.069) | -.907 (.050) | -.984 (.045) | -.961 (.045) | -.089 (.116) | -.067 (.092) | -.533 (.109) | -.519 (.093) | -.807 (.068) | -.874 (.067) | -.889 (.049) | -.911 (.044) | -.948 (.044) | .315 (.13) | .204 (.103) | -.130 (.121) | -.296 (.104) | -.593 (.076) | -.676 (.075) | -.833 (.055) | -.907 (.049) | -.870 (.049) | .225 (.119) | .016 (.094) | -.411 (.111) | -.496 (.095) | -.740 (.069) | -.814 (.069) | -.837 (.050) | -.899 (.045) | -.907 (.045) | .135 (.087) | .093 (.069) | -.447 (.082) | -.489 (.070) | -.768 (.051) | -.768 (.051) | -.808 (.037) | -.865 (.033) | -.882 (.033) | -.010 (.096) | .035 (.076) | -.384 (.090) | -.455 (.077) | -.707 (.056) | -.753 (.056) | -.818 (.040) | -.904 (.036) | -.889 (.036) | .116 (.090) | .120 (.071) | -.404 (.084) | -.467 (.072) | -.769 (.053) | -.787 (.052) | -.867 (.038) | -.911 (.034) | -.889 (.034) | .171 (.087) | .142 (.069) | -.383 (.081) | -.475 (.070) | -.737 (.051) | -.737 (.050) | -.871 (.037) | -.942 (.033) | -.954 (.033)
Statistical Analysis 1: Comparison: Stress, Immediate, Males, CS+ vs Stress, Immediate, Males, GS1 vs Stress, Immediate, Males, GS2 vs Stress, Immediate, Males, GS3 vs Stress, Immediate, Males, GS4 vs Stress, Immediate, Males, GS5 vs Stress, Immediate, Males, GS6 vs Stress, Immediate, Males, GS7 vs Stress, Immediate, Males, CS- vs Stress, Delayed, Males, CS+ vs Stress, Delayed, Males, GS1 vs Stress, Delayed, Males, GS2 vs Stress, Delayed, Males, GS3 vs Stress, Delayed, Males, GS4 vs Stress, Delayed, Males, GS5 vs Stress, Delayed, Males, GS6 vs Stress, Delayed, Males, GS7 vs Stress, Delayed, Males, CS- vs Sham Control, Immediate, Males, CS+ vs Sham Control, Immediate, Males, GS1 vs Sham Control, Immediate, Males, GS2 vs Sham Control, Immediate, Males, GS3 vs Sham Control, Immediate, Males, GS4 vs Sham Control, Immediate, Males, GS5 vs Sham Control, Immediate, Males, GS6 vs Sham Control, Immediate, Males, GS7 vs Sham Control, Immediate, Males, CS- vs Sham Control, Delayed, Males, CS+ vs Sham Control, Delayed, Males, GS1 vs Sham Control, Delayed, Males, GS2 vs Sham Control, Delayed, Males, GS3 vs Sham Control, Delayed, Males, GS4 vs Sham Control, Delayed, Males, GS5 vs Sham Control, Delayed, Males, GS6 vs Sham Control, Delayed, Males, GS7 vs Sham Control, Delayed, Males, CS- vs Stress, Immediate, Females, CS+ vs Stress, Immediate, Females, GS1 vs Stress, Immediate, Females, GS2 vs Stress, Immediate, Females, GS3 vs Stress, Immediate, Females, GS4 vs Stress, Immediate, Females, GS5 vs Stress, Immediate, Females, GS6 vs Stress, Immediate, Females, GS7 vs Stress, Immediate, Females, CS- vs Stress, Delayed, Females, CS+ vs Stress, Delayed, Females, GS1 vs Stress, Delayed, Females, GS2 vs Stress, Delayed, Females, GS3 vs Stress, Delayed, Females, GS4 vs Stress, Delayed, Females, GS5 vs Stress, Delayed, Females, GS6 vs Stress, Delayed, Females, GS7 vs Stress, Delayed, Females, CS- vs Sham Control, Immediate, Females, CS+ vs Sham Control, Immediate, Females, GS1 vs Sham Control, Immediate, Females, GS2 vs Sham Control, Immediate, Females, GS3 vs Sham Control, Immediate, Females, GS4 vs Sham Control, Immediate, Females, GS5 vs Sham Control, Immediate, Females, GS6 vs Sham Control, Immediate, Females, GS7 vs Sham Control, Immediate, Females, CS- vs Sham Control, Delayed, Females, CS+ vs Sham Control, Delayed, Females, GS1 vs Sham Control, Delayed, Females, GS2 vs Sham Control, Delayed, Females, GS3 vs Sham Control, Delayed, Females, GS4 vs Sham Control, Delayed, Females, GS5 vs Sham Control, Delayed, Females, GS6 vs Sham Control, Delayed, Females, GS7 vs Sham Control, Delayed, Females, CS-; Test type: Superiority; p = 0.998, ANOVA

7. Secondary Outcome: Change in Baseline Salivary Cortisol (Nmol/l)
Description: Saliva samples were collected from participants prior to undergoing the stress or sham control condition (baseline) and then 25 min later. The change in salivary cortisol levels was analyzed. Greater levels indicated greater cortisol responses to stress.
Time Frame: Day 1 (change from baseline to 25 min post-stress)
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some salivary cortisol levels were unable to be obtained due to a lack of adequate saliva.
Measure: Mean (Standard Error); unit: Change in cortisol (nmol/l)
Groups:
- Stress, Immediate, Males: Change in salivary cortisol levels on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males: Change in salivary cortisol levels on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males: Change in salivary cortisol levels on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Change in salivary cortisol levels on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Change in salivary cortisol levels on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Change in salivary cortisol levels on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Change in salivary cortisol levels on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Change in salivary cortisol levels on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 41 | 39 | 35 | 38 | 75 | 60 | 73 | 78
Change in cortisol (nmol/l) | 1.413 (.308) | 1.014 (.315) | -.039 (.333) | .236 (.320) | .728 (.227) | .710 (.254) | .558 (.231) | -.091 (.223)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.10, ANOVA

8. Secondary Outcome: Change in Baseline Salivary Alpha-amylase (U/ml)
Description: Saliva samples were collected from participants prior to undergoing the stress or sham control condition (baseline) and then immediately after the manipulation. The change in salivary alpha-amylase levels was analyzed. Greater levels indicated greater alpha-amylase responses to stress.
Time Frame: Day 1 (change from baseline to immediately after stress)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Change in alpha-amylase (U/ml)
Groups:
- Stress, Immediate, Males: Change in salivary alpha-amylase levels on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males: Change in salivary alpha-amylase levels on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males: Change in salivary alpha-amylase levels on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Change in salivary alpha-amylase levels on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Change in salivary alpha-amylase levels on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Change in salivary alpha-amylase levels on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Change in salivary alpha-amylase levels on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Change in salivary alpha-amylase levels on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 39 | 40 | 35 | 43 | 68 | 55 | 70 | 73
Change in alpha-amylase (U/ml) | 4.210 (7.132) | -12.943 (7.042) | 7.656 (7.528) | -3.411 (6.792) | 17.561 (5.40) | 2.608 (6.005) | 5.090 (5.323) | -3.601 (5.213)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.992, ANOVA

9. Secondary Outcome: Average Subjective Pain, as Assessed by Verbal Self Report
Description: During the stress or sham control manipulation, participants rated the painfulness of the water bath at 1-minute intervals on an 11-point scale ranging from 0-10, with 0 = lack of pain and 10 = unbearable pain. The obtained ratings were averaged and analyzed. Greater ratings indicated greater subjective pain during the stressor.
Time Frame: Stress or sham control condition on Day 1
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some participants did not report subjective pain ratings.
Measure: Mean (Standard Error); unit: score on a scale of 0-10
Groups:
- Stress, Immediate, Males: Average pain ratings on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males: Average pain ratings on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average pain ratings on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average pain ratings on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average pain ratings on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Average pain ratings on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average pain ratings on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average pain ratings on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on a scale of 0-10 | 6.089 (.228) | 6.415 (.223) | .123 (.243) | .159 (.226) | 6.806 (.167) | 6.765 (.181) | .092 (.172) | .131 (.163)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.519, ANOVA

10. Secondary Outcome: Average Subjective Stress, as Assessed by Verbal Self Report
Description: During the stress or sham control manipulation, participants rated the stressfulness of the water bath at 1-minute intervals on an 11-point scale ranging from 0-10, with 0 = lack of stress and 10 = unbearable stress. The obtained ratings were averaged and analyzed. Greater ratings indicated greater subjective stress during the stressor.
Time Frame: Stress or sham control condition on Day 1
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some participants did not report subjective stress ratings.
Measure: Mean (Standard Error); unit: score on scale of 0-10
Groups:
- Stress, Immediate, Males: Average stress ratings on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males: Average stress ratings on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average stress ratings on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average stress ratings on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average stress ratings on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Average stress ratings on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average stress ratings on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average stress ratings on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on scale of 0-10 | 4.457 (.289) | 5.778 (.283) | .675 (.307) | .318 (.286) | 5.910 (.212) | 5.843 (.230) | .184 (.217) | .405 (.207)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.007, ANOVA

11. Secondary Outcome: Change in Heart Rate (Bpm)
Description: Heart rate (bpm) measurements were aken via the PPG module of the Biopac MP150 system from participants prior to undergoing the stress or sham control condition (baseline) and then halfway through the manipulation.The change in heart rate was analyzed.
Time Frame: Day 1 (change from baseline to during stress or sham control manipulation)
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some heart rate measurements were unable to be obtained from participants due to technical issues (e.g., pulse oximeter malfunction).
Measure: Mean (Standard Error); unit: Change in heart rate (beats per minute)
Groups:
- Stress, Immediate, Males: Change in heart rate on Day 1 in males stressed immediately before learning
- Stress, Delayed, Males: Change in heart rate on Day 1 in males stressed 30 min before learning
- Sham Control, Immediate, Males: Change in heart rate on Day 1 in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Change in heart rate on Day 1 in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Change in heart rate on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Change in heart rate on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Change in heart rate on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Change in heart rate on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 42 | 45 | 37 | 43 | 78 | 67 | 74 | 81
Change in heart rate (beats per minute) | 4.924 (1.159) | 3.922 (1.120) | -.379 (1.235) | .345 (1.146) | 5.339 (.851) | 4.348 (.918) | .096 (.873) | -1.337 (.835)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.457, ANOVA

12. Secondary Outcome: Change in Salivary Progesterone (pg/ml)
Description: Saliva samples were collected from female participants prior to undergoing the stress or sham control condition (baseline) and then 25 min later. The change in salivary progesterone levels were analyzed.
Time Frame: Day 1 (change from baseline to 25 min post-stress)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Change in progesterone (pg/ml)
Groups:
- Stress, Immediate, Females: Change in salivary progesterone levels on Day 1 in females stressed immediately before learning
- Stress, Delayed, Females: Change in salivary progesterone levels on Day 1 in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Change in salivary progesterone levels on Day 1 in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Change in salivary progesterone levels on Day 1 in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 64 | 52 | 60 | 61
Change in progesterone (pg/ml) | 247.165 (51.177) | 160.933 (56.776) | 197.625 (52.856) | 198.469 (52.421)
Statistical Analysis 1: Comparison: Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.415, ANOVA

13. Other Pre Specified Outcome: Salivary Estradiol (pg/ml)
Description: Salivary estradiol (pg/ml) was measured by enzyme immunoassay (Salimetrics LLC) performed on saliva samples collected from female participants on Days 1 and 2.
Time Frame: Average across Day 1 (baseline) and Day 2 (baseline)
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Stress, Immediate, Females: Average estradiol levels in females stressed immediately before learning
- Stress, Delayed, Females: Average estradiol levels in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average estradiol levels in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average estradiol levels in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 79 | 66 | 73 | 78
pg/ml | 2.040 (.131) | 2.050 (.144) | 1.971 (.137) | 1.955 (.132)
Statistical Analysis 1: Comparison: Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.923, ANOVA

14. Other Pre Specified Outcome: State Anxiety
Description: The Spielberger State-Trait Anxiety Inventory (STAI) was administered following generalization testing on Day 2. The STAI provides scores (20-80) for state and trait anxiety. State anxiety was used for this measure and was a sum of 20 items from the STAI. The minimum score for state anxiety was 20, and the maximum score was 80. Higher scores represented higher levels of state anxiety.
Time Frame: Day 2 - following generalization testing
Population: The overall number of participants analyzed is not consistent with the numbers in the participant flow module. Some participants did not complete the questionnaire.
Measure: Mean (Standard Error); unit: score on a scale of 20-80
Groups:
- Stress, Immediate, Males: Average state anxiety in males stressed immediately before learning
- Stress, Delayed, Males: Average state anxiety in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average state anxiety in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average state anxiety in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average state anxiety in females stressed immediately before learning
- Stress, Delayed, Females: Average state anxiety in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average state anxiety in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average state anxiety in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on a scale of 20-80 | 38.395 (1.738) | 36.422 (1.699) | 37.868 (1.849) | 38.750 (1.718) | 43.213 (1.274) | 41.441 (1.382) | 40.868 (1.307) | 41.845 (1.244)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.981, ANOVA

15. Other Pre Specified Outcome: Childhood Trauma Questionnaire (CTQ)
Description: The Childhood Trauma Questionnaire (CTQ) was administered following generalization testing on Day 2. The questionnaire consists of 25 items and yields a score between 25 and 125. Higher scores represent greater levels of childhood trauma exposure.
Time Frame: Day 2 - following generalization testing
Population: as for outcome 14
Measure: Mean (Standard Error); unit: score on a scale of 25-125
Groups:
- Stress, Immediate, Males: Total CTQ score in males stressed immediately before learning
- Stress, Delayed, Males: Total CTQ score in males stressed 30 min before learning
- Sham Control, Immediate, Males: Total CTQ score in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Total CTQ score in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Total CTQ score in females stressed immediately before learning
- Stress, Delayed, Females: Total CTQ score in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Total CTQ score in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Total CTQ score in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on a scale of 25-125 | 34.93 (1.836) | 32.600 (1.795) | 31.632 (1.953) | 34.909 (1.815) | 37.688 (1.346) | 34.471 (1.460) | 35.184 (1.381) | 35.333 (1.314)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.627, ANOVA

16. Other Pre Specified Outcome: Anxiety Sensitivity Index
Description: The Anxiety Sensitivity Index (ASI) was administered following generalization testing on Day 2. The ASI consists of 18 items and yields a score that reflects an individual's dispositional anxiety sensitivity. The minimum score is 0, and the maximum score is 72. Greater scores reflect a greater sensitivity to anxiety.
Time Frame: Day 2 - following generalization testing
Population: as for outcome 14
Measure: Mean (Standard Error); unit: score on a scale of 0-72
Groups:
- Stress, Immediate, Males: Average anxiety sensitivity in males stressed immediately before learning
- Stress, Delayed, Males: Average anxiety sensitivity in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average anxiety sensitivity in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average anxiety sensitivity in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average anxiety sensitivity in females stressed immediately before learning
- Stress, Delayed, Females: Average anxiety sensitivity in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average anxiety sensitivity in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average anxiety sensitivity in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on a scale of 0-72 | 16.047 (1.649) | 15.933 (1.612) | 14.816 (1.754) | 14.591 (1.630) | 18.838 (1.209) | 16.882 (1.311) | 17.171 (1.240) | 15.619 (1.180)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.901, ANOVA

17. Other Pre Specified Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: The Center for Epidemiological Studies Depression Scale (CES-D) was administered following generalization testing on Day 2. The CES-D is a 20-item measure of symptoms of depression. The possible range for scores is 0-60 with higher scores suggesting more severe symptoms of depression.
Time Frame: Day 2 - following generalization testing
Population: as for outcome 14
Measure: Mean (Standard Error); unit: score of a scale of 0-60
Groups:
- Stress, Immediate, Males: Average CES-D score in males stressed immediately before learning
- Stress, Delayed, Males: Average CES-D score in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average CES-D score in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average CES-D score in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average CES-D score in females stressed immediately before learning
- Stress, Delayed, Females: Average CES-D score in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average CES-D score in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average CES-D score in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score of a scale of 0-60 | 12.767 (1.439) | 10.000 (1.407) | 15.579 (1.531) | 10.909 (1.423) | 15.950 (1.055) | 13.441 (1.144) | 13.974 (1.082) | 14.583 (1.030)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.166, ANOVA

18. Other Pre Specified Outcome: PTSD Checklist - Civilian Version
Description: The PTSD Checklist - Civilian Version was administered following generalization testing on Day 2. The checklist is a 17-item measure of symptoms of post-traumatic stress disorder (PTSD). The minimum score is 0, and the maximum score is 80. Greater scores reflect greater symptoms related to PTSD.
Time Frame: Day 2 - following generalization testing
Population: as for outcome 14
Measure: Mean (Standard Error); unit: score on a scale of 0-80
Groups:
- Stress, Immediate, Males: Average PTSD score in males stressed immediately before learning
- Stress, Delayed, Males: Average PTSD score in males stressed 30 min before learning
- Sham Control, Immediate, Males: Average PTSD score in males exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Males: Average PTSD score in males exposed to the sham manipulation 30 min before learning
- Stress, Immediate, Females: Average PTSD score in females stressed immediately before learning
- Stress, Delayed, Females: Average PTSD score in females exposed to stress 30 min before learning
- Sham Control, Immediate, Females: Average PTSD score in females exposed to the sham manipulation immediately before learning
- Sham Control, Delayed, Females: Average PTSD score in females exposed to the sham manipulation 30 min before learning
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
Number analyzed (Participants) | 43 | 45 | 38 | 44 | 80 | 68 | 76 | 84
score on a scale of 0-80 | 31.628 (1.774) | 29.800 (1.734) | 34.868 (1.887) | 30.886 (1.754) | 36.088 (1.301) | 32.456 (1.411) | 34.868 (1.335) | 34.190 (1.269)
Statistical Analysis 1: Comparison: Stress, Immediate, Males vs Stress, Delayed, Males vs Sham Control, Immediate, Males vs Sham Control, Delayed, Males vs Stress, Immediate, Females vs Stress, Delayed, Females vs Sham Control, Immediate, Females vs Sham Control, Delayed, Females; Test type: Superiority; p = 0.252, ANOVA

ADVERSE EVENTS:
Time Frame: 2 days, the length of the time of in-person experimental sessions
Arm/Group | Stress, Immediate, Males | Stress, Delayed, Males | Sham Control, Immediate, Males | Sham Control, Delayed, Males | Stress, Immediate, Females | Stress, Delayed, Females | Sham Control, Immediate, Females | Sham Control, Delayed, Females
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/59 | 0/58 | 0/57 | 0/97 | 0/87 | 0/94 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/59 | 0/58 | 0/57 | 0/97 | 0/87 | 0/94 | 0/98
Other Adverse Events (participants affected / at risk) | 0/56 | 0/59 | 0/58 | 0/57 | 0/97 | 0/87 | 0/94 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03786952/Prot_SAP_ICF_000.pdf